CLINICAL TRIAL: NCT00405210
Title: Open-label, Multicenter,PhaseI Trial in Order To Determine the Safety and Pharmacokinetics of BAY43-9006 in Combination With Docetaxel as First-line Treatment in Metastatic Hormone Refractory Prostate Cancer Patients
Brief Title: Pharmacokinetic Study of BAY43-9006 and Taxotere to Treat Patient With Prostatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Cliniques universitaires Saint-Luc-Université Catholique de Louvain, Prof. J-P Machiels
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL-ONCO 06-003; BAY 43-9006/12180
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Primary Disease; Prostate Cancer
Keywords: hormone-resistant; metastatic prostatic cancer; pharmacokinetics; naïve patient
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sorafenib; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sorafenib (200 or 400mg bid) and taxotere iv — 200 mg BID, day 3-19 cycle 1, day 2-19 other cycles 200 mg BID, day 3-21 Cycle 1, day 1-21 other cycles 400 mg BID, day 3-19 cycle 1, day 2-19 other cycles 400 mg BID, day 3-21 cycle 1, day 1-21 other cycles
  Other Names: Nexavar

SUMMARY:
The purpose of the trial is to determine the most effective dose of BAy 46-9003 associated to taxotere for first-line treatment of patient with prostatic cancer.

BAY 43-9006 (SORAFENIB) is a novel dual-action Raf kinase and VEGFR inhibitor, which is orally available and has a favorable safety profile in patients with advanced solid tumors. This, together with the antitumor activity observed after treatment with BAY 43-9006 (SORAFENIB), provides a rationale for further evaluation in patients with advanced cancer. The recommended dose of BAY 43-9006 (SORAFENIB) for future studies is 400 mg bid as a continuous dosing schedule.

DETAILED DESCRIPTION:
This study propose to treat patients with metastatic and hormone-refractory prostatic cancer in first intention. There is no limits of age from 18 years old. A new inhibitor of angiogenesis (Sorafenib) is associated to the standard treatment in this type of pathology.

Patients have to demonstrate radiologically a disease progression and also a progression based on increase of psa level.

The main objective is to Determine the recommended dose of BAY 43-9006 in combination with docetaxel in hormone-refractory prostate cancer patients as first line treatment in patients with metastatic hormone-refractory prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to beginning protocol specific procedures.
* 18 years
* Radiologically proven presence of metastases
* Histologically/cytologically proven prostate adenocarcinoma.
* Biochemically evaluable disease
* Patients must have received prior hormonal therapy as defined below:

  * Castration by orchiectomy and/or LHRH agonists with or without
  * Antiandrogens
  * Other hormonal agents (e.g., ketoconazole, ...)
* The testosterone level should be < 50 ng/dl (10) documented disease progression defined by PSA increase. Patients must have a value of at least 5 ng/ml in addition to increasing PSA to be eligible.
* Life expectancy > 3 months
* ECOG performance status 0-2.
* Normal cardiac function.

Exclusion Criteria:

* Prior chemotherapy except estramustine phosphate.
* Prior isotope therapy (e.g., strontium, samarium).
* Prior radiotherapy to >25% of bone marrow
* Prior therapy with anti-VEGF therapy
* Prior malignancy except the following: adequately treated basal cell or squamous cell skin cancer, or any other cancer from which the patient has been disease-free for >5 years.
* History or presence of central nervous system (CNS) disease (i.e. primary brain tumor, malignant seizures, CNS metastases or carcinomatous meningitis)
* Symptomatic peripheral neuropathy
* Other serious illness or medical condition the use of corticosteroids.
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational drug within 30 days prior to study screening.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BAY 9006.
* Major surgery with 4 weeks of study entry
* Autologous bone marrow transplant or stem cell rescue within 4 months of study entry
* Use of biologic response modifiers, such as G-CSF, within 3 weeks of study entry
* Treatment with any other anti-cancer therapy (except LHRH agonists) including any prescribed compounds and/or OTC products for the treatment of prostate cancer must be stopped.
* Treatment with drugs that are metabolized by the cytochrome P450 system (i.e warfarin sodium,…)
* Treatment with systemic corticosteroids used for reasons other than specified by the protocol must be stopped.
* Biphosphonates could not be initiated after inclusion into the protocol. At inclusion, patients receiving biphosphonates with a PSA progression could continue biphosphonates.
* Patients with reproductive potential not employing an effective method of birth control. Barrier contraceptives must be used throughout the trial.
* Inadequate recovery from previous surgery, radiation, chemo-, biologic or immunotherapy
* Patients who have known hypersensitivity to the study medication
* Substance abuse, medical social, psychological conditions that may interfere with the subject's participation in the study or evaluation of study results
* Patients unable to sallow oral medications.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-09; Primary Completion 2008-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Determine the recommended dose of BAY 43-9006 (SORAFENIB) in combination with docetaxel in hormone-refractory prostate cancer patients as first line treatment in patients with metastatic hormone refractory prostate cancer. | after the first 24 patients

SECONDARY OUTCOMES:
Evaluation of pharmacokinetics and pharmacodynamics of BAY43-9006 in combination with docetaxel* | after the first 24 patients
Toxicity and safety | at end of study
Response rate in patients with measurable disease | at end of study
PSA response rate | at end of study
PSA response duration | at end of study
Time to PSA progression (=time between treatment start and PSA progression) | at end of study
Time to PSA progression after the last dose of docetaxel in patients with no progression after stopping docetaxel (= time between the last dose of docetaxel and PSA progression) | at end of study
Event progression-free survival | at end of study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal H Machiels, Prof, Study Director — Cliniques Universitaires St Luc -UCL
Locations (6):
- Belgium (5):
  - St Pierre, Ottignies, Brabant Wallon
  - Cliniques Universitaires St Luc, Brussels, Brussels Capital
  - Notre Dame et Reine Fabiola, Charleroi, Hainaut
  - Sainte Elisabeth, Namur, Namur
  - Clinique Universiataire de Mont Godinne, Yvoir, Namur
- Hôpital Européen Georges Pompidou, Paris, France